CLINICAL TRIAL: NCT01755364
Title: A Trial to Assess the Immunogenicity and Safety of the Trivalent Virosomal Influenza Vaccine, Formulation of 2012-2013, in Healthy Subjects Aged Over 3 Years Old to 18 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLUV12T13C
Record Dates: First submitted 2012-12-17; First posted 2012-12-24 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdimFlu-V (Experimental)
  Interventions: Biological: AdimFlu-V

INTERVENTIONS:
Biological: AdimFlu-V

SUMMARY:
This is an open study of the use of AdimFlu-V (2012-2013 season) vaccine in young healthy subjects. Subjects aged equal to or over 9 years old and less than 18 years old will receive one dose of vaccine (0.5 mL) by intramuscular injection into the upper arm. Subjects aged equal to or over 3 years old and less than 9 years old will received two doses of vaccine (0.5 mL) by intramuscular injection into the upper arm separated by 4 weeks (28 days). Safety outcomes included immediate reactions at the time of vaccination, solicited local and systemic reactions within 7 days after each vaccination, unsolicited adverse events observed since first vaccination to 28 days after the last dose of vaccination, and serious adverse events during the observation. Sera prepared from blood samples will be collected from each subject immediately prior to, and 4 weeks after each vaccination. Anti-hemagglutinin (HA) antibody titers will be determined using the WHO hemagglutination inhibition reference technique. The central laboratory who is responsible for antibody titrations will not be aware of the background of blood samples (e.g., pre- or post-serum), it is also called observer-blinded. All subjects will be followed, either by clinical visit or by telephone contact, for 8 weeks after the last vaccination for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Boys or non-pregnant girls and aged ≥ 3 through < 18 years old on the day of first vaccination;
2. Subject and/or parents(s)/legal guardian(s) must be willing to comply with planned study procedures and be available for all study visits;
3. Subject must be in good physical health on the basis of medical history, physical examination;
4. Subject and/or parents(s)/legal guardian(s) must provide the signed study-specific informed consent prior to initiation of any study procedure.

Exclusion Criteria:

1. Subjects received influenza vaccine within the previous 6 months;
2. History of hypersensitivity to eggs or hen's protein, polymyxin B, or neomycin, or similar pharmacological effects to study vaccine;
3. Personal or family history of Guillain-Barré Syndrome;
4. An acute febrile illness within 1 week prior to vaccination;
5. Current upper respiratory illness, including the common cold or nasal congestion within 72 hours;
6. Subjects with influenza-like illness as defined by the presence of fever (temperature ≥ 38°C) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
7. Female subjects who are pregnant, lactating or likely to become pregnant during the study; women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study;
8. Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before study vaccination;
9. Immunodeficiency, or under immunosuppressive treatment;
10. Receipt of live virus vaccine within 1 month prior to study vaccination or expect receipt within 1 month of study vaccination; receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt within 1 month of study vaccination;
11. Receipt of any blood products, including immunoglobulin in the prior 3 months;
12. Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine;
13. Significant chronic illness for which inactivated influenza vaccine is recommended or commonly used.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2013-01-28 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the immunogenicity profiles for influenza virus vaccine strains (2012-2013 season) of the AdimFlu-V. | Change from baseline for anti-hemaglutinin (HA) antibodies by hemagglutinaton inhibition (HAI) at 28 days post immunization
  Serum samples will be obtained prior to vaccination, and 4 weeks post each vaccination. Serum samples will be tested for anti-hemagglutinin (HA) antibodies by hemagglutination inhibition (HAI) and assays will be performed at Adimmune Corporation designated central laboratory. Subjects will be considered to be seronegative if serum HAI titer < 1:10. The seroconversion is defined as the post-vaccination serum HAI titer at least 1:40 for whom had negative pre-vaccination or a four-fold or greater increase in HAI titers in subjects who had positive pre-vaccination serum.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-V. | 7 days of each vaccination and 8 weeks after last vaccination
  Reactogenicity events are pre-specified adverse events systematically recorded on diary cards (a grid of check boxes for each event and each day) during the immediate post-vaccination period by all participants. In general, reactogenicity events will be recorded for 7 days after each vaccination. The selection of the events to be collected systematically is based on events expected to occur with wild-type influenza infection including fever (≥38°C), runny nose or nasal congestion, cough, sore throat, muscle aches, headache, vomiting, nausea and malaise. Furthermore, the local (injection site) reactions will also be evaluated that include soreness/pain, swelling, redness, ecchymosis and limitation of arm motion.
  In regard to the long term safety of the study vaccine, the significant and/or serious adverse event(s) will be recorded during the 8 weeks follow up after the scheduled last vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Linkuo, Taoyuan District, Taiwan